CLINICAL TRIAL: NCT07033598
Title: A Randomized Phase 2 Study of Pacritinib vs. Hydroxyurea in Patients With Advanced Proliferative Chronic Myelomonocytic Leukemia
Brief Title: Pacritinib vs. Hydroxyurea in Advanced Proliferative Chronic Myelomonocytic Leukemia
Acronym: PROSPERA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Theradex (Industry)
Collaborators: MDS/MPN International Working Group (UK Sponsor) (Unknown); Sobi, Inc. (Industry); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROSPERA; ABNL-MARRO 002 (Other: MDS/MPN International Working Group (IWG))
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by prior therapy. Within each stratum, participants will be randomly assigned to receive either pacritinib or hydroxyurea in a 2:1 ratio.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pacritinib (Experimental): Pacritinib 200 mg twice daily
  Interventions: Drug: Pacritinib
- Hydroxyurea (Active Comparator): Hydroxyurea at doses up to 4 g daily
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Pacritinib — 100-mg capsules
  Arms: Pacritinib
Drug: Hydroxyurea — capsules or tablets
  Arms: Hydroxyurea

SUMMARY:
The goal of this clinical trial is to learn if pacritinib works better than hydroxyurea to treat advanced proliferative chronic myelomonocytic leukemia in adults. The main questions it aims to answer are:

* Does pacritinib improve disease control compared to hydroxyurea?
* What medical problems do participants have when taking pacritinib or hydroxyurea? Researchers will compare pacritinib to hydroxyurea to see if pacritinib is more effective and better tolerated in people with advanced proliferative chronic myelomonocytic leukemia.

Participants will be randomly assigned to receive either pacritinib twice a day or hydroxyurea for up to 48 weeks.

After treatment ends, participants will be followed for up to one year.

DETAILED DESCRIPTION:
This is a randomized, multicenter, open-label Phase 2 clinical trial evaluating the efficacy and safety of pacritinib compared to hydroxyurea in adult participants with advanced proliferative chronic myelomonocytic leukemia (CMML). Approximately 66 participants will be randomized in a 2:1 ratio to receive either pacritinib 200 mg twice daily (n=44) or hydroxyurea (n=22) for up to 48 weeks. Randomization will be stratified based on prior therapy (i.e., prior use of hydroxyurea or hypomethylating agents vs. no prior therapy).

The study includes:

* A 28-day screening period
* A 48-week treatment period
* A 30-day post-treatment follow-up
* A survival follow-up phase lasting approximately one year after randomization Participants receiving pacritinib who are not deriving benefit by Week 24, as assessed by the treating physician, will discontinue treatment. Participants in the hydroxyurea arm who are not deriving benefit by Week 24-or who experience non-leukemic disease progression-may switch to pacritinib for the remainder of the treatment period, provided they meet predefined "Safe to Switch" criteria.

Participants who discontinue study therapy due to toxicity, disease progression, or other protocol-defined criteria will enter survival follow-up to monitor overall survival, event-free survival, leukemic-free survival, and receipt of allogeneic hematopoietic stem cell transplant. Data will be collected at least every three months until death, hematopoietic stem cell transplant, or leukemic transformation.

An independent data monitoring committee will oversee safety, with the first review after enrollment of ~18 participants and subsequent reviews approximately every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CMML-1 (5th WHO classification), with <10% bone marrow blasts on morphology and <5% peripheral blood blasts.
* Proliferative disease, defined as white blood cell count ≥13 × 10⁹/L.
* Advanced disease, defined as at least one of the following features during screening: spleen palpable ≥5cm below the lower costal margin in the midclavicular line; TSS ≥20; or platelet count <100 × 10⁹/L. For participants in whom spleen palpation is not feasible, an ultrasound exam may be performed for assessment of spleen craniocaudal length (length ≥12 cm by ultrasound is considered splenomegaly).
* ECOG performance status ≤2.
* Adequate organ function: AST and ALT ≤3 × ULN, total bilirubin ≤4 × ULN (≤8 × ULN in participants with Gilbert's syndrome), creatinine clearance >30 mL/min, absolute neutrophil count ≥0.5 × 10⁹/L, PT and PTT ≤1.5 × ULN.
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and, along with male participants, must agree to use a highly effective method of contraception from the first dose through 90 days after the last dose.

Exclusion Criteria:

* Active malignancy diagnosed within the past 2 years, except for curatively treated non-invasive cancers (e.g., basal/squamous cell skin cancer, low-risk prostate cancer on stable endocrine therapy with PSA stable ≥3 months).
* Allogeneic hematopoietic stem cell transplant within 12 months prior to enrollment, or requiring immunosuppressive therapy within 6 months before enrollment.
* Likely to undergo allogeneic hematopoietic stem cell transplant within 6 months, per investigator assessment.
* Prior systemic treatment with any JAK inhibitor.
* Treatment with hypomethylating agents or cytotoxic chemotherapy (excluding hydroxyurea) within 28 days prior to enrollment.
* Participation in another interventional study or use of experimental therapy within 28 days or 5 half-lives, whichever is longer.
* Use of hematologic support drugs within 28 days prior to enrollment. Supportive care permitted.
* Use of strong CYP3A4 inhibitors or inducers within 14 days or 5 half-lives before enrollment, whichever is shorter.
* Use of systemic anticoagulants or antiplatelets (except aspirin ≤100 mg/day) within 14 days prior. Therapeutic anticoagulation allowed if stable for ≥90 days without bleeding events.
* CTCAE Grade ≥2 bleeding within 3 months prior to enrollment, unless due to a reversible cause (e.g., trauma, surgery).
* QTcF >450 ms (men) or >470 ms (women); QTcF up to 480 ms allowed if QRS >100 ms. QTcF may be repeated if affected by reversible factors.
* CTCAE Grade ≥3 cardiac event within 3 months before enrollment.
* Symptomatic heart failure with limitations on ordinary activity.
* Uncontrolled infection at study entry.
* Moderate/severe hepatic impairment (Child-Pugh B or C), or active viral hepatitis:
* HBV: Exclude if HBsAg+ or HBV DNA detectable. HBV antiviral therapy allowed if HBV DNA undetectable.
* HCV: Allowed if HCV Ab+ but RNA negative.
* Uncontrolled HIV or detectable viral load while on antiretrovirals.
* Known hypersensitivity to pacritinib or its excipients (microcrystalline cellulose, polyethylene glycol, magnesium stearate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit at Week 24, defined as achieving erythroid response in the absence of leukemic transformation. | Measured from Week 24 through the end of treatment, up to 48 weeks.
  For participants with baseline hemoglobin <10 g/dL, response is defined as either a ≥1.5 g/dL hemoglobin increase lasting ≥8 weeks without red blood cell transfusion, or, if transfusion-dependent at baseline (≥4 units in the 8 weeks pre-enrollment), achieving ≥8 weeks of red blood cell transfusion independence, excluding transfusions given for pretreatment Hb ≤8.5 g/dL.
  Leukemic transformation is defined as ≥20% blasts or blast equivalents in the peripheral blood or bone marrow biopsy, or development of granulocytic sarcoma.
Clinical benefit at Week 24, defined as achieving platelet response in the absence of leukemic transformation. | Measured from Week 24 through the end of treatment, up to 48 weeks.
  For participants with baseline platelet counts <100 × 10⁹/L, response is defined as one of the following: an increase to ≥20 × 10⁹/L and by ≥100% for ≥8 weeks without platelet transfusion (if baseline <20 × 10⁹/L); an increase of ≥30 × 10⁹/L for ≥8 weeks without transfusion (if baseline 20-<100 × 10⁹/L); or, if transfusion-dependent at baseline (≥4 units in the 8 weeks pre-enrollment), achieving ≥8 weeks of platelet transfusion independence.
  Leukemic transformation is defined as ≥20% blasts or blast equivalents in the peripheral blood or bone marrow biopsy, or development of granulocytic sarcoma.
Clinical benefit at Week 24, defined as achieving neutrophil response in the absence of leukemic transformation. | Measured from Week 24 through the end of treatment, up to 48 weeks.
  For participants with baseline ANC ≤1 × 10⁹/L, response is defined as either an increase to >0.5 × 10⁹/L and by ≥100% for ≥8 weeks without myeloid growth factors (if baseline ANC ≤0.5 × 10⁹/L), or an increase by ≥50% for ≥8 weeks without myeloid growth factors (if baseline ANC >0.5 to ≤1 × 10⁹/L).
  Leukemic transformation is defined as ≥20% blasts or blast equivalents in the peripheral blood or bone marrow biopsy, or development of granulocytic sarcoma.
Clinical benefit at Week 24, defined as achieving spleen response in the absence of leukemic transformation. | Measured from Week 24 through the end of treatment, up to 48 weeks.
  For participants with baseline spleen ≥5 cm below the left costal margin (midclavicular line), spleen response is defined as a ≥35% reduction in spleen volume at endpoint assessment by MRI or CT.
  Leukemic transformation is defined as ≥20% blasts or blast equivalents in the peripheral blood or bone marrow biopsy, or development of granulocytic sarcoma.
Clinical benefit at Week 24, defined as achieving symptom response in the absence of leukemic transformation. | Measured from Week 24 through the end of treatment, up to 48 weeks.
  Among participants with baseline Total Symptom Score (TSS) ≥20 per the MPN-SAF TSS: achieving ≥50% TSS reduction from baseline at the time of endpoint assessment.
  Leukemic transformation is defined as ≥20% blasts or blast equivalents in the peripheral blood or bone marrow biopsy, or development of granulocytic sarcoma.

SECONDARY OUTCOMES:
Clinical benefit at any time, defined as achieving at least one of the primary endpoint clinical benefit response criteria at any time on study. | Measured from the start of study treatment to the end of treatment, for up to 48 weeks.
Achieving response at Week 24 and 48 according to the IWG 2015 criteria), including the following subtypes: complete response, complete cytogenetic remission, partial remission, marrow response | Measured from Week 24 through the end of treatment, up to 48 weeks.
Duration of response for primary endpoint (clinical benefit by Week 24) | Measured from Week 24 through the end of treatment, up to 48 weeks.
Event-free survival | Measured from the start of study treatment to the end of treatment, for up to 48 weeks.
  Event-free survival is defined as the time without death from any cause, transformation to AML (including granulocytic sarcoma), or disease progression after ≥3 cycles (Week 12), including CMML-1 to CMML-2 with ≥5% absolute blast increase or worsening splenomegaly.
Leukemia-free survival, where events include death from any cause or transformation to AML (including granulocytic sarcoma) | Measured from the start of study treatment to the end of treatment, for up to 48 weeks.
Overall survival | Measured from the date of initiating study treatment to the date of death from any cause, assessed up to 24 months.
Incidence of allogeneic hematopoietic stem cell transplant. | Measured from the date of initiating study treatment to the date of allogeneic hematopoietic stem cell transplant., assessed for up to 24 months
Adverse events and laboratory abnormalities as graded by NCI CTCAE v5.0. | From the start of the adverse event collection period through 30 days following the last dose of study treatment.
Change in arterial blood pressure measured in mmHg. | From the start of the study treatment through 30 days following the last dose of study treatment.
Change in pulse rate measured in beats per minute. | From the start of the study treatment through 30 days following the last dose of study treatment.
Change in respiratory rate measured in breaths per minute. | From the start of the study treatment through 30 days following the last dose of study treatment.
Change in corrected QT interval measured in milliseconds using 12-lead electrocardiogram. | From the start of the study treatment through 30 days following the last dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States